CLINICAL TRIAL: NCT00990795
Title: A Randomized Trial of Cyclosporine for Myocardial Protection During Open Heart Surgery
Brief Title: Trial of Cyclosporine for Myocardial Protection During Open Heart Surgery
Acronym: CYCLO1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Jon-Cecil Walkes, MD, University of Texas Medical School Houston
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYCLO1
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Cardiac Surgical Procedures
Keywords: open heart surgery; cyclosporine; myocardial protection
MeSH Terms: interventions — Cyclosporine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine (Experimental): Cyclosporine Group: Patients will receive a dose of cyclosporine just after they are heparinized. They will receive 2.5 mg of cyclosporine (Sandimmune, Novartis) per kilogram of body weight. It will be injected into a central venous line at the time the central venous line is inserted by the anesthesia team.
  Interventions: Drug: cyclosporine
- Placebo (Placebo Comparator): Placebo: Patients will undergo the cardiac surgery procedures using standard technique. They will have ischemic arrest of the heart with cold blood cardioplegia using standardized methods of myocardial protection or off-pump CABG. The patients in the placebo group will receive a volumetrically equivalent dose of normal saline to the cyclosporine dose.
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: cyclosporine — Cyclosporine Patients will receive a dose of cyclosporine just after they are heparinized. They will receive 2.5 mg of cyclosporine (Sandimmune, Novartis) per kilogram of body weight. It will be injected into a central venous line at the time the central venous line is inserted by the anesthesia team.
  Arms: Cyclosporine
Drug: saline solution — Placebo Group: Patients will undergo the cardiac surgery procedures using standard technique. They will have ischemic arrest of the heart with cold blood cardioplegia using standardized methods of myocardial protection or off-pump CABG. The patients in the placebo group will receive a volumetrically equivalent dose of normal saline to the cyclosporine dose.
  Arms: Placebo

SUMMARY:
Administration of cyclosporine has been found to have a myocardial protective effect, improving post-operative cardiac function in patients undergoing percutaneous coronary interventions by diminishing infarct size. The purpose of the proposed study is to conduct a randomized, controlled clinical trial in patients undergoing isolated valvular heart surgery, or coronary artery bypass surgery. Specifically the investigators will evaluate the cardio-protective effects of cyclosporine on post ischemic-arrest myocardium. The two factors will be treatment group and cyclosporine versus placebo.

DETAILED DESCRIPTION:
The specific aim of this study is to perform a randomized controlled study to compare the effects of cyclosporine v. placebo on changes in myocardial functioning associated with open heart surgery for isolated valvular or coronary artery bypass procedures.

The research question is:

Compared to placebo, does administration of cyclosporine just before surgery improve myocardial functioning in terms of:

* Transthoracic ECHO (TTE) assessment of ejection fraction
* Cardiac index (CI), mixed venous oxygen saturation (SVO2), systemic vascular resistance (SVR)
* Length of stay
* 30-d mortality
* Angina Scale
* SF-36 measure of quality of life
* Measures associated with myocardial function:

  1. Cardiac Index
  2. Blood glucose level
  3. Serum Troponin I level
  4. Free Fatty Acid levels
  5. Serum CPK-MB levels
  6. Serum phosphoratase levels

ELIGIBILITY:
Inclusion criteria:

* Men and women, 18 years of age or older
* Patients with multi-vessel coronary artery disease
* Patients undergoing isolated valvular heart surgery (aortic/ mitral)
* Patients undergoing CABG

Exclusion Criteria:

* Patients with cardiac arrest
* Patients with ventricular fibrillation
* Patients with cardiogenic shock
* Patients requiring circulatory arrest
* Patients with known hypersensitivity to cyclosporine
* Patients with known renal failure or a GFR <50 ml/min/1.732
* Patients with liver failure
* Patients with uncontrolled hypertension
* Women who are pregnant or who are of childbearing age and not on contraception
* Patients with a serum bilirubin level greater than 3 mg/100 mL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Length of Stay (LOS) | postoperative to 30 days

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (TTE) | postoperative
Cardiac Index | postoperative
SVO2 | Postoperative
Systemic Vascular Resistance (SVR) | postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jon-Cecil M Walkes, MD, Principal Investigator — University of Texas Medical School Houston; Heinrich Taegtmeyer, MD, Study Director — University of Texas Medical School Houston; George K Goodrick, PhD, Study Chair — University of Texas Medical School Houston
Locations (1):
- University of Texas Medical School Houston, Houston, Texas, United States